CLINICAL TRIAL: NCT07243067
Title: Tumor-Derived Extracellular Vesicles for Noninvasive Molecular Classification of Kidney Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 25-003121; HT9425-25-1-0607 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2025-11-14; First posted 2025-11-21 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Renal Cell Carcinoma; Clear-cell Renal Cell Carcinoma; Papillary Renal Cell Carcinoma; Chromophobe Renal Cell Carcinoma; Kidney Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Clear-cell RCC: Participants with clear-cell RCC
  Interventions: Other: Proteomic profiling of urinary EVs; Procedure: Blood sample collection
- Papillary RCC: Participants with papillary RCC
  Interventions: Other: Proteomic profiling of urinary EVs; Procedure: Blood sample collection
- Chromophobe RCC: Participants with chromophobe RCC
  Interventions: Other: Proteomic profiling of urinary EVs; Procedure: Blood sample collection
- Benign Renal Tumor: Participants with benign renal tumors
  Interventions: Other: Proteomic profiling of urinary EVs

INTERVENTIONS:
Other: Proteomic profiling of urinary EVs — EV isolation and mass spectrometry.
Procedure: Blood sample collection — Blood samples collected pre- and post-nephrectomy
  Groups: Chromophobe RCC; Clear-cell RCC; Papillary RCC

SUMMARY:
This is a correlative (lab-based) study aiming to identify protein markers in urine extracellular vesicles (EVs) that can be used to develop non-invasive molecular tests for patients with renal cell carcinoma (RCC). Aim 1 will use urine collected previously in biorepository. Aim 2 will prospectively collect blood specimens pre and post nephrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Urine sample in existing biorepository
* High-risk renal cell carcinoma (RCC) per American Urological Association (AUA) guidelines
* Scheduled to undergo nephrectomy

Exclusion Criteria:

* Does not meet inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Mayo Clinic patients scheduled to undergo nephrectomy for treatment of RCC.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Differentiate tumor-derived extracellular vesicle (tdEV) surface proteins expressed in benign vs malignant renal tumors | Baseline
  Differential protein expression analysis will be performed on stored urine samples from a biorepository to identify tdEV proteins in each renal cell carcinoma (RCC) subtype (clear-cell, papillary, and chromophobe) versus benign.
Prediction of metastasis after surgery | Perioperative (pre- and post-nephrectomy),
  Blood samples will be collected pre-and post-nephrectomy to asses for tdEV levels which will be correlated with clinicopathological features to test whether tdEV levels can be used to better predict likelihood of metastasis in patients undergoing curative-intent radical nephrectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Lucien-Matteoni, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No